CLINICAL TRIAL: NCT06378593
Title: An Open-Label, Multi-center Phase 1/2 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Activity of 3HP-2827 in Patients With Unresectable or Metastatic Solid Tumors With FGFR2 Alterations
Brief Title: A Study of 3HP-2827 in Treatment of Unresectable or Metastatic Solid Tumors With FGFR2 Alterations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 3H (Suzhou) Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3HP-2827-102
Record Dates: First submitted 2024-03-29; First posted 2024-04-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors With FGFR2 Alterations, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage I - dose escalation (Experimental): Dose escalation of 3HP-2827 in patients with advanced solid tumors.
  Interventions: Drug: 3HP-2827
- Stage II - expansion (Experimental): Expansion evaluating the recommended dose and schedule of 3HP-2827 identified from Stage I.
  Interventions: Drug: 3HP-2827

INTERVENTIONS:
Drug: 3HP-2827 — 3HP-2827 will be administered orally once daily in 28-day cycles.

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of 3HP-2827 in the treatment of unresectable or metastatic solid tumors with FGFR2 alterations.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to provide written informed consent and has the ability to comply with the study protocol
* Men or women, age ≥ 18 years at the time of signing informed consent.
* Histologically or cytologically confirmed surgically unresectable, locally advanced, metastatic solid tumor.
* ECOG score is 0 or 1.
* An expected survival of ≥ 12 weeks.
* Evaluable or measurable disease per RECIST v1.1.
* Adequate organ function, as measured by laboratory values.

Exclusion Criteria:

* Active brain metastases.
* Have other malignancies within the past 3 years.
* The toxicity from previous anti-tumor treatment has not recovered to ≤ grade 1.
* Clinically significant corneal or retinal disease/keratopathy.
* Clinically significant cardiovascular disorders.
* Failure to swallow, chronic diarrhea, or presence of other factors affecting drug absorption.
* Known to be allergic to any study drug or any of its excipients.
* Assessed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2028-06-16 (Estimated); Study Completion 2028-06-16 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Stage- incidence of adverse events (AEs) | From baseline up until 28 days after the final dose
Dose Escalation Stage- incidence of dose-limiting toxicities (DLTs) | Days 1-28 of Cycle 1 (a cycle is 28 days)
Dose Escalation Stage -Percentage of Participants With Changes From Baseline in Targeted Vital Signs | From baseline up until 28 days after the final dose
Dose Escalation Stage -Percentage of Participants With Changes From Baseline in Targeted Clinical Laboratory Test Results | From baseline up until 28 days after the final dose
Dose Escalation Stage -Percentage of Participants With Changes From Baseline in Targeted ECG Parameters | From baseline up until 28 days after the final dose
Dose Escalation Stage -determine the maximum tolerated dose (MTD) and/or the recommended dose (RD) for expansion stage or recommended Phase II dose (RP2D) of 3HP-2827 | Initiation of study drug until study discontinuation, (up to approximately 24 months)
Expansion stage -Objective response rate（ORR） | Initiation of study drug until disease progression (up to approximately 36 months)
  ORR refers to the percentage of patients with best overall response of confirmed CR or PR from the start of study treatment to patient withdrawal due to PD.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) during the dosing interval of 3HP-2827 and/or its major metabolites as monotherapy. | Initiation of study drug until study discontinuation, (up to approximately 24 months))
Time to maximum concentration (Tmax) of 3HP-2827 and/or its major metabolites as monotherapy. | Initiation of study drug until study discontinuation, (up to approximately 24 months))
Apparent clearance (CL/F) of 3HP-2827 and/or its major metabolites as monotherapy. | Initiation of study drug until study discontinuation, (up to approximately 24 months))
Area under the concentration-time curve (AUC) of 3HP-2827 and/or its major metabolites as monotherapy. | Initiation of study drug until study discontinuation, (up to approximately 24 months))
Terminal half life (t1/2) of 3HP-2827 and/or its major metabolites as monotherapy. | Initiation of study drug until study discontinuation, (up to approximately 24 months))
Apparent volume of distribution (Vz/F) of 3HP-2827 and/or its major metabolites as monotherapy. | Initiation of study drug until study discontinuation, (up to approximately 24 months))
Duration of Response (DOR) as assessed by RECIST v1.1 | Up to 45 months
  DOR refers to the time period from the first evaluation of confirmed CR or PR (whichever occurs first) to PD or death.
Disease control rate (DCR) as assessed by RECIST v1.1 | Up to 45 months
  DCR refers to the percentage of patients with best overall response of confirmed CR, PR or SD from the start of study treatment to patient withdrawal due to PD.
Progression-free survival (PFS) as assessed by RECIST v1.1 | Up to 45 months
  PFS refers to the time between the date of first dose and the first PD or death due to any cause based on the investigator's imaging review results
Overall survival (OS) | Up to 48 months
  OS refers to the time from the date of first dose to the date of death due to any cause.
Dose escalation stage - Objective Response Rate (ORR) | Up to 45 months
  ORR refers to the percentage of patients with best overall response of confirmed CR or PR from the start of study treatment to patient withdrawal due to PD.
Expansion Stage- incidence of adverse events (AEs) | From baseline up until 28 days after the final dose
Expansion Stage -Percentage of Participants With Changes From Baseline in Targeted Vital Signs | From baseline up until 28 days after the final dose
Expansion Stage -Percentage of Participants With Changes From Baseline in Targeted Clinical Laboratory Test Results | From baseline up until 28 days after the final dose
Expansion Stage -Percentage of Participants With Changes From Baseline in Targeted ECG Parameters | From baseline up until 28 days after the final dose
Expansion Stage -Changes in patient-reported outcomes as assessed by the European Organization for Research and Treatment of Cancer Core QoL Questionnaire (EORTC QLQ-C30) in patients with advanced solid tumors | From baseline up until 28 days after the final dose

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - ZhongShan Hospital, Shanghai, Shanghai Municipality